CLINICAL TRIAL: NCT06013618
Title: Clinical Analysis of Naxitamab (hu3F8) in the Treatment of Pediatric High Risk or Refractory/ Relapsed Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hainan General Hospital (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director, Sun Yat-sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3F8-RWS
Record Dates: First submitted 2023-08-19; First posted 2023-08-28 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Irinotecan; Topoisomerase I Inhibitors; Temozolomide; Injections; Combined Modality Therapy; sintilimab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- naxitamab and GM-CSF only (Other): Suitable for patients with high risk neuroblastoma who obtain CR after chemotherapy combined with surgery, radiotherapy and/or hematopoietic stem cell transplantation. The treatment cycle is repeated every 4 weeks for a total of 5 courses, and discontinuation of nasetuzumab and GM-CSF should be considered if disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Naxitamab monotherapy; Drug: GM-CSF
- naxitamab and GM-CSF in combination with irinotecan and temozolomide (Other): Suitable for high-risk group neuroblastoma treated by chemotherapy combined with surgery, radiotherapy and or hematopoietic stem cell transplantation patients with tumor residual or progression during treatment (refractory); Patients who relapse after initial treatment. Repeat every 3 weeks until tumor progression, patient withdrawal, or toxicity becomes intolerable, up to 8 procedures.
  Interventions: Drug: Irinotecan; Drug: Temozolomide; Drug: Naxitamab in combination therapy; Drug: GM-CSF with combination regimen
- naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody (Other): Suitable for high-risk group neuroblastoma treated by chemotherapy combined with surgery, radiotherapy and or hematopoietic stem cell transplantation patients with tumor residual or progression during treatment (refractory); Patients who relapse after initial treatment. Repeat every 3 weeks until tumor progression, patient withdrawal, or toxicity becomes intolerable, up to 8 procedures.
  Interventions: Drug: Irinotecan; Drug: Temozolomide; Drug: Naxitamab in combination therapy; Drug: GM-CSF with combination regimen; Drug: Sintilimab

INTERVENTIONS:
Drug: Naxitamab monotherapy — Naxitamab is administered on days 1, 3, and 5
  Other Names: hu3F8
  Arms: naxitamab and GM-CSF only
Drug: GM-CSF — Each treatment cycle is 28 days and is started with five days (days -4 to 0) of GM-CSF administered at 250 mcg/m2/day in advance of the start of naxitamab infusion. GM-CSF is thereafter administered at 500 mcg/m2/day on days 1 to 5.
  Other Names: Recombinant Human Granulocyte/Macrophage Colony-stimulating Factor
  Arms: naxitamab and GM-CSF only
Drug: Irinotecan — Each HITS treatment cycle is 21 days. Irinotecan intravenously (IV) at 50 mg/m2/day will be administered from Day 1-5 concurrently with temozolomide orally at 150 mg/m2/day or 100 mg/m2/day.
  Other Names: DNA topoisomerase I inhibitor
  Arms: naxitamab and GM-CSF in combination with irinotecan and temozolomide; naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody
Drug: Temozolomide — Each HITS treatment cycle is 21 days. Irinotecan intravenously (IV) at 50 mg/m2/day will be administered from Day 1-5 concurrently with temozolomide orally at 150 mg/m2/day or 100 mg/m2/day.
  Other Names: Temozolomide for Injection
  Arms: naxitamab and GM-CSF in combination with irinotecan and temozolomide; naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody
Drug: Naxitamab in combination therapy — Naxitamab 2.25mg/kg IV will be administered on Days 2, 4, 8 and 10.
  Other Names: hu3F8
  Arms: naxitamab and GM-CSF in combination with irinotecan and temozolomide; naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody
Drug: GM-CSF with combination regimen — GM-CSF 250 mcg/m2/day will be administered subcutaneously on Days 6-10.
  Other Names: Recombinant Human Granulocyte/Macrophage Colony-stimulating Factor
  Arms: naxitamab and GM-CSF in combination with irinotecan and temozolomide; naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody
Drug: Sintilimab — Sintilimab was administerd with 3mg/kg (max 200mg) on day 11 every 3 weeks.
  Other Names: PD-1 antibody
  Arms: naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody

SUMMARY:
This is an prospective study to evaluate the safety and efficacy of naxitamab monotherapy or combined with chemotherapy or combined with chemotherapy and checkpoint inhibitor in the treatment of pediatric high-risk and refractory/relapsed neuroblastoma in Sun Yat-sen University Cancer Center.

DETAILED DESCRIPTION:
Patients with high risk neuroblastoma who obtain CR after chemotherapy combined with surgery, radiotherapy and/or hematopoietic stem cell transplantation received axitamab and GM-CSF. Patients with high-risk neuroblastoma treated by chemotherapy combined with surgery, radiotherapy and or hematopoietic stem cell transplantation patients with tumor residual or progression during treatment (refractory) received naxitamab and GM-CSF in combination with irinotecan and temozolomide or naxitamab and GM-CSF in combination with irinotecan and temozolomide and PD-1 antibody.

ELIGIBILITY:
Inclusion Criteria:

1)Confirmed diagnosis of high-risk NB 2)1 year of age or above 3)Patient or parent/guardian must provide written informed consent to participate 4)If patient is sexually active, the patient agrees to use effective contraception 5)Confirmed negative urine pregnancy test for sexually active female of child-bearing potential (post-menarche)

Exclusion Criteria:

1. Significant organ toxicity
2. Known or suspected allergy or hypersensitivity to anti-GD2 antibodies or to GM-CSF or its s components.
3. Patient is pregnant, planning to become pregnant (while being treated with naxitamab) or is currently breastfeeding
4. Patient will undergo treatment with another investigational drug, whilst being treated with naxitamab or has received another investigational drug within the 4 weeks prior to commencing treatment with naxitamab
5. Patient is either eligible and able to participate in or is currently participating in an active interventional Y-mAbs sponsored clinical trial with naxitamab within the indication applied for
6. Patient is unable to comply with the naxitamab treatment or has a medical condition that would potentially increase the severity of the toxicities experienced from naxitamab treatment at the discretion of the treating physician
7. Left ventricular ejection fraction of <50% by echocardiography OR other clinically relevant cardiac disorders at the discretion of the investigator
8. Inadequate pulmonary function defined as evidence of dyspnea at rest, exercise intolerance, and/or chronic oxygen requirement. In addition, room air pulse oximetry < 94% and/or abnormal pulmonary function tests if these assessments are clinically indicated

   Applicable for treatment with naxitamab in combination with GM-CSF only:
9. Patient has active progression of the NB disease
10. Patient has active NB disease at primary site or soft-tissue metastasis
11. Patient has known CNS metastases when initiating naxitamab treatment

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | from start of naxitamab treatment to 1.5 years after EOT
  The proportion of patients who achieved CR or PR

SECONDARY OUTCOMES:
DCR | from start of naxitamab treatment to 1.5 years after EOT
  The proportion of patients who achieved CR or PR or SD
EFS | from start of naxitamab treatment to 1.5 years after EOT
  The time from from start of naxitamab treatment to disease progression, recurrence
OS | from start of naxitamab treatment to 1.5 years after EOT
  The time from from start of naxitamab treatment to death or loss of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Study Chair — SunYat Sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No